CLINICAL TRIAL: NCT00235456
Title: Supplemental Perioperative Oxygen Reduces the Risk of Surgical Wound Infection: A Randomized, Double-blind Trial
Brief Title: Supplemental Oxygen Reduces Surgical Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Professor & Chair, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RETIQ
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Wound Infection
Keywords: oxygen; surgical complications; colo-rectal resections
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 80% perioperative oxygen (Active Comparator): Perioperative supplemental oxygen: Patients were randomly assigned to 80% fraction of inspired oxygen (FIO2) intraoperatively and for 6 hours after surgery. Anesthetic treatment and antibiotic administration were standardized.
  Interventions: Procedure: Perioperative supplemental oxygen
- 30% perioperative oxygen (Placebo Comparator): Standard oxygen: Patients were randomly assigned to 30% fraction of inspired oxygen (FIO2) intraoperatively and for 6 hours after surgery. Anesthetic treatment and antibiotic administration were standardized.
  Interventions: Procedure: Standard oxygen

INTERVENTIONS:
Procedure: Perioperative supplemental oxygen — Patients were assigned to 80% fraction of inspired oxygen (FIO2) intraoperatively and for 6 hours after surgery. Anesthetic treatment and antibiotic administration were standardized.
  Arms: 80% perioperative oxygen
Procedure: Standard oxygen — Patients were assigned to 30% fraction of inspired oxygen (FIO2) intraoperatively and for 6 hours after surgery. Anesthetic treatment and antibiotic administration were standardized.
  Arms: 30% perioperative oxygen

SUMMARY:
Supplemental perioperative oxygen has been reported to halve or double the risk of surgical wound infection. We tested the hypothesis that supplemental oxygen reduces infection risk following colorectal surgery. Colorectal surgery patients (n=300) were randomly assigned to 30% or 80% FiO2 intraoperatively and 6 hours postoperatively. Wound infections were diagnosed by blinded investigators using Centers for Disease Control criteria. Baseline patient characteristics, anesthetic management, and potential confounding factors were recorded. Wound infection rates were compared with chi-square analysis. Logistic regression identified the contribution of potential confounding factors. Surgical wound infection occurred in 24.4% of patients receiving 30% oxygen, but only 14.9% of those receiving 80% oxygen (P<0.039). According to logistic regression, the relative risk of infection in patients given supplemental oxygen was 0.46 (P=0.035). Supplemental inspired oxygen reduced wound infection risk by roughly a factor of two. We thus recommend that supplemental oxygen be provided to patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Context: Supplemental perioperative oxygen has been variously reported to halve or double the risk of surgical wound infection.

Objective: We tested the hypothesis that supplemental oxygen reduces infection risk following colorectal surgery.

Design: Randomized, controlled trial. Setting: Fourteen Spanish hospitals. Patients: Three hundred patients undergoing elective colorectal surgery. Interventions: Patients were randomly assigned to either 30% or 80% FiO2 intraoperatively and for 6 hours after surgery. Anesthetic management and antibiotic administration were standardized.

Main outcome measures: Wound infections were diagnosed by blinded investigators using Centers for Disease Control criteria. Baseline patient characteristics, anesthetic management, and potential confounding factors were recorded. The wound infection rate in the 30% and 80% oxygen groups was compared with chi-square analysis. A logistic regression was used to identify the contribution of potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal resection,
* Patients having abdominal-peritoneal reconstructions were included, but not those scheduled for minor colon surgery (e.g., polypectomy, isolated colostomy) or laparoscopic surgery.

Exclusion Criteria:

* Exclusion criteria included expected surgery time of less than one hour, fever or existing signs of infection, diabetes mellitus (type I or II), HIV infection, weight loss exceeding 20% in the previous three months, serum albumin concentration < 30 g/L, and a leukocyte count <2500 cells/ml.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-03; Primary Completion 2004-10 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Javier Belda, MD, PhD, Study Director — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico Universitario, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belda FJ, Aguilera L, Garcia de la Asuncion J, Alberti J, Vicente R, Ferrandiz L, Rodriguez R, Company R, Sessler DI, Aguilar G, Botello SG, Orti R; Spanish Reduccion de la Tasa de Infeccion Quirurgica Group. Supplemental perioperative oxygen and the risk of surgical wound infection: a randomized controlled trial. JAMA. 2005 Oct 26;294(16):2035-42. doi: 10.1001/jama.294.16.2035. PMID 16249417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Started | 150 | 150
Completed | 148 | 143
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen | Total
Number analyzed (Participants) | 148 | 143 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.8) | 62.3 (12.5) | 63.3 (12.2)
Gender [Count of Participants; unit: Participants]
  Female | 77 | 52 | 129
  Male | 71 | 91 | 162

OUTCOME MEASURES:

1. Primary Outcome: Incisional Surgical Wound Infection
Description: Surgical wounds were defined as infected if they met Centers for Disease Control and Prevention definitions.
Time Frame: 0 to 14 days after surgery
Measure: Number; unit: participants
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
participants | 22 | 35
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.04, Chi-squared; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.38 to 0.98]

2. Secondary Outcome: Return of Bowel Function
Description: Time to return of bowel function, measured in days.
Time Frame: time to event after surgery to discharge from hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
days | 3 (1.5) | 3.1 (1.7)
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.54, t-test, 2 sided

3. Secondary Outcome: Return to Ambulation
Description: time to return to ambulation after surgery, measured in days
Time Frame: time to event after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
days | 3.9 (2.2) | 4.2 (2.6)
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.28, t-test, 2 sided

4. Secondary Outcome: First Solid Food Intake
Description: Time to restarting feeding after surgery, measured in days.
Time Frame: time to event after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
days | 4.2 (2.2) | 4.4 (2.0)
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.57, t-test, 2 sided

5. Secondary Outcome: Staples Removed
Description: Time to staples removed, measured in days
Time Frame: time to event after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
days | 10.5 (3.3) | 10.3 (3.0)
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.71, t-test, 2 sided

6. Secondary Outcome: Hospital Length of Stay
Description: The number of days patient stayed in the hospital after surgery.
Time Frame: time to hospital discharge after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Number analyzed (Participants) | 148 | 143
days | 11.7 (7) | 10.5 (4.4)
Statistical Analysis 1: Comparison: 80% Perioperative Oxygen vs 30% Perioperative Oxygen; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | 80% Perioperative Oxygen | 30% Perioperative Oxygen
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/143
Other Adverse Events (participants affected / at risk) | 0/148 | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No